CLINICAL TRIAL: NCT03816280
Title: Cerebrovascular Effects of the Use of Alpha-stat or pH-stat Management of Cardiopulmonary Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Collaborators: GINOP (Unknown); Hungarian Basic Research Council (Other)
Responsible Party: Principal Investigator, Barna Babik, Professor, Szeged University
Other Study IDs: WHO2788-b
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Cardiac Surgical Procedures
Keywords: Spectroscopy, Near-Infrared
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group T2DM-alpha: Patients with diabetes mellitus undergoing CPB with alpha-stat acid-base management
  Interventions: Procedure: Elective cardiopulmonary bypass (CPB); Procedure: Alpha-stat acid-base management
- Group T2DM-pH: Patients with diabetes mellitus undergoing CPB with pH-stat acid-base management
  Interventions: Procedure: Elective cardiopulmonary bypass (CPB); Procedure: pH-stat acid-base management
- Group Ctrl-alpha: Control patients undergoing CPB with alpha-stat acid-base management
  Interventions: Procedure: Elective cardiopulmonary bypass (CPB); Procedure: Alpha-stat acid-base management
- Group Ctrl-pH: Control patients undergoing CPB with pH-stat acid-base management
  Interventions: Procedure: Elective cardiopulmonary bypass (CPB); Procedure: pH-stat acid-base management

INTERVENTIONS:
Procedure: Elective cardiopulmonary bypass (CPB) — All groups undergo elective cardiopulmonary bypass (CPB)
Procedure: Alpha-stat acid-base management — Acid-base status during CPB will be maintained using the alpha-stat regime
  Groups: Group Ctrl-alpha; Group T2DM-alpha
Procedure: pH-stat acid-base management — Acid-base status during CPB will be maintained using the pH-stat regime
  Groups: Group Ctrl-pH; Group T2DM-pH

SUMMARY:
Type 2 diabetes mellitus (T2DM) poses a significant burden on the patients and the health care system. The increasing number of surgery performed in elderly population results in an increased number of perioperative T2DM-related adverse effects. T2DM has a prevalence of 30-40% in a population undergoing cardiovascular surgery. Cardiac surgery, especially cardiopulmonary bypass (CPB) is also known to deteriorate cerebral oxygenation.

Furthermore, acid-base balance of patients undergoing CPB can be managed using two main regimes: alpha-stat and pH-stat. The use of pH-stat acid-base management involves maintaining the patient's temperature-corrected pH at a constant level (7.40) and maintaining normocapnia (pCO2 of 40 mmHg). Alpha-stat acid-base management on the other hand is performed by maintaining the ionization state of histidine by keeping the pH stable when a standardized temperature of 37C is used. Therefore, while a constant pH (7.40) and normocapnia (pCO2 of 40 mmHg) are targeted when measured at 37C, the hypothermia applied during CPB will result in a lower pCO2 and in a relative respiratory alkalosis. Previous studies investigating alpha-stat and pH-stat managements demonstrated increased jugular venous oxygen concentrations when pH-stat management was applied.

Therefore, our study is aimed at characterizing the effects of an alpha-stat or pH-stat acid-base management regime on the cerebral oxygenation, parameters of regional cerebral oxygen supply and demand during and following CPB in diabetic patients. These parameters include regional cerebral tissue oxygen saturation (rSO2), central venous oxygen saturation ScvO2) and the physiological saturation gap between ScvO2 and rSO2 (gSO2).

DETAILED DESCRIPTION:
One hour before the surgery, patients are premedicated with lorazepam (per os, 2.5 mg). Induction of anaesthesia is achieved by iv midazolam (30 μg/kg), sufentanyl (0.4-0.5 μg/kg), and propofol (0.3-0.5 mg/kg), and iv propofol (50 mg/kg/min) is administered to maintain anaesthesia. Intravenous boluses of rocuronium (0.6 mg/kg for induction and 0.2 mg/kg every 30 minutes for maintenance) is administered iv to ensure neuromuscular blockade. A cuffed tracheal tube (internal diameter of 7, 8, or 9 mm) is used for tracheal intubation, and patients are mechanically ventilated (Dräger Zeus, Lübeck, Germany) in volume-controlled mode with decelerating flow. A tidal volume of 7 ml/kg and a positive end-expiratory pressure of 4 cmH2O are applied, and the ventilation frequency is adjusted to 12-14 breaths/min to maintain end-tidal CO2 partial pressure of 36 38 mmHg. Mechanical ventilation is performed with a fraction of inspired oxygen of 0.5 before CPB, and it is increased to 0.8 after CPB. As a standard part of the cardiac anaesthesia procedure, oesophageal and rectal temperature probes are introduced, and a central venous line is inserted into the right jugular vein. The left radial artery is also cannulated to monitor systolic, diastolic and mean arterial (MAP) blood pressures and arterial blood gas samples.

The membrane oxygenator is primed with 1,500 ml lactated Ringer's solution prior to CPB. Intravenous heparin (300 U/kg) is injected into the patient, to achieve an activated clotting time of 400 s during CPB procedures. During CPB, mild hypothermia is allowed, the mechanical ventilation is stopped, and the ventilator is disconnected without applying positive airway pressure. Before restoring ventilation, the lungs are inflated 3-5 times to a peak airway pressure of 30 cmH2O to facilitate lung recruitment.

After securing arterial and peripheral venous lines and placement of NIRS and entropy sensors, data collection is initiated immediately before anesthesia induction in all groups of patients. Since catheterization of the jugular vein is scheduled after anesthesia induction, ScvO2 and gSO2 data are not available at the first protocol stage. After induction and before surgical incision, all measurements are repeated. The whole data set is registered at the beginning of CPB after clamping the aorta and 5 min before the end of CPB. The final stage of the protocol is allocated to the end of the operation after sternal closure. All invasive (i.e. arterial and venous blood gas) and non-invasive (i.e. NIRS) data are registered simultaneously at each protocol stage.

Sample sizes are estimated to enable the detection of a 10% difference in the primary outcome parameter gSO2 that we considered clinically significant. Accordingly, sample-size estimation based on an ANOVA test with 4 groups of patients (diabetic and control patients undergoing CPB with alpha-stat or pH-stat acid-base regime) indicated that 100 patients were required in each group to detect a significant difference between the protocol groups.

Two-way repeated measures ANOVA with the inclusion of an interaction term is used for all measured variables with the protocol stage as within-subject factor (protocol stages) and group allocation as between-subject factor to establish the effects of T2DM and the acid-base management regime on the parameters of cerebral oxygenation. At half-way of the data collection, an interim analyses will be performed and the further data collection will be proceeded based on the results of this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with or without diabetes mellitus
* age between 18-80 years

Exclusion Criteria:

* patients older than 80 years of age
* poor ejection fraction (<40%)
* unilateral internal carotid stenosis (>75%)
* medical history of smoking
* medical history of chronic obstructive pulmonary disease
* medical history of stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled at the Second Department of Internal Medicine and Cardiology Centre Cardiac Surgical Unit, University of Szeged
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation | Intraoperative interval during cardiac surgery starting from anaesthesia induction until end of the surgery. (approx. 180 minutes, measurements at ~0-40-140-160 minutes).
  The spatially resolved continuous-wave NIRS technique is applied to estimate cerebral tissue oxygen saturation. This monitor uses two different wavelengths (730 and 810 nm) and has two detectors positioned 3 and 4 cm from the light source. Computing the differences between the intensity of the emitted and the reflected light with two receivers allows the measurement of the oxygen saturation of the cerebral cortex. In this study, two adult sensors are applied on the left and right sides of the patient's forehead symmetrically, and the cerebral-tissue oxygen saturation is monitored continuously during the surgical procedures and the data are registered in each protocol stage. The mean value of the rSO2 measured by the sensors is calculated for each protocol stage and used for further analyses.
Central venous oxygen saturation | Intraoperative interval during cardiac surgery starting from anaesthesia induction until end of the surgery. (approx. 180 minutes, measurements at ~0-40-140-160 minutes).
  The central venous oxygen saturation is measured from central venous blood samples (Radiometer ABL 505, Copenhagen, Denmark). The proper positioning of the central venous catheter is verified by the surgeon via manually palpating the catheter tip.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Centre Cardiac Surgical Unit and Second Department of Internal Medicine, University of Szeged, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: Undecided